CLINICAL TRIAL: NCT03237650
Title: Conditioned Pain Modulation Using Painful Cutaneous Electrical Stimulation or Simply Habituation?
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med., Ruhr University of Bochum
Other Study IDs: PCES-Hab
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Habituation
Keywords: Painful cutaneous electrical stimulation; Conditioned Pain Modulation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Painful cutaneous electrical stimulation (PCES) and corresponding evoked potentials led to a significant pain relief and decrease of evoked potentials and has been used to analyze conditioned pain modulation (CPM). However, it is unknown whether the pain relief results from habituation to the repeated painful electric stimulation. We compared the effects of CPM and habituation on PCES-induced pain and PCES-evoked potentials and analyzed whether increased attention by a random change of electric intensities amplifies the habituation effects.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any kind of disease

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
pain relief | during the measurement
  pain intensity of painful cutaneous electrical stimulation on a numeric rating scale (NRS 0-100)
N1P1-amplitude | during the measurement
  Amplitudes of painful cutaneous electrical stimulation evoked potentials in µV

SECONDARY OUTCOMES:
N1-latency | during the measurement
  Latency of the peak N1 of painful cutaneous electrical stimulation evoked potentials in msec
P0N1-amplitude | during the measurement
  Amplitudes of painful cutaneous electrical stimulation evoked potentials in µV

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof Dr med, Principal Investigator — University clinic Bergmannsheil Bochum gGmbH, Department of pain medicine

IPD SHARING:
Plan to Share IPD: No